CLINICAL TRIAL: NCT00581269
Title: Dietary Intervention and Exercise Training (DIET) in Moderate to Severe Chronic Kidney Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: the Fellow conducting the study left the institution in 2009
Sponsor: Vanderbilt University (Other)
Responsible Party: Alp Ikizler, MD, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 070990
Record Dates: First submitted 2007-12-18; First posted 2007-12-27 (Estimated); Last update posted 2010-11-03 (Estimated); Status verified 2010-11

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Diet, Fat-Restricted; Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): low-impact aerobic exercise group
  Interventions: Behavioral: low-impact aerobic exercise
- 2 (Active Comparator): dietary restriction group
  Interventions: Dietary Supplement: low-calorie (low-fat) diet
- 3 (No Intervention): control group

INTERVENTIONS:
Behavioral: low-impact aerobic exercise — subjects will undergo supervised physical activity for a maximum of 30-60 minutes, every other day, 3 days per week for 3 months; to offer variety in the exercise prescription, subjects will alternately use a treadmill, an elliptical trainer, a Nu-Step cross-trainer and a recumbent stationary bicycle
  Arms: 1
Dietary Supplement: low-calorie (low-fat) diet — subjects will undergo a 20% reduction in total daily calories from their usual daily energy consumption every day for 3 months
  Arms: 2

SUMMARY:
The oxidative stress and inflammatory state is known to contribute to the pathogenesis of atherosclerosis, and is predictive of cardiovascular events and mortality rates in the general population and patients with chronic kidney disease (CKD), particularly in patients with end stage renal disease (ESRD) on dialysis therapy 1. Increased oxidative stress and inflammation has been identified in all stages of CKD, ranging from moderate renal insufficiency to ESRD. However, the pathophysiology of increased oxidative stress and inflammation associated with the development of CKD is currently poorly understood.

There is also concern about the epidemic of obesity in the United States, as the overall health status of the general population is adversely affected by increasing adiposity. Recent studies indicate a strong relationship between adiposity and incident CKD. Furthermore, the presence of an elevated body mass index (BMI) is an independent predictor for progression to ESRD, even after additional adjustments for baseline blood pressure and the presence or absence of diabetes mellitus. Limited data in the general population show that healthy lifestyle interventions, such as exercise and dietary caloric restriction, either alone or in combination, reduce the inflammatory and oxidative stress burden seen in obese subjects. The impact of healthy lifestyle modifications on inflammation and oxidative stress has not been investigated in the obese CKD population. Based on the foregoing observations, the purpose of this investigation will be to determine whether healthy lifestyle interventions in the form of low-impact aerobic exercise and dietary calorie restriction in obese subjects (BMI ≥ 30kg/m2) with moderate to severe (Stage III-IV) CKD [estimated glomerular filtration rate (GFR) 20-59 ml/min] will improve oxidative stress, inflammation, insulin resistance, adipocytokines, endothelial dysfunction, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Stage III-IV (estimated GFR 20-59 min/ml) chronic kidney disease measured by MDRD formula.
2. BMI ≥ 30 kg/m2
3. Age > 18 or < 65 years.
4. Life expectancy greater than one year.
5. Ability to understand and provide informed consent for participation in the study.

Exclusion Criteria:

1. Active inflammatory disease such as: AIDS (HIV seropositivity is not an exclusion criteria), active hepatitis C or B, active gout, other active inflammatory diseases.
2. Active malignancy excluding basal or squamous cell carcinoma of the skin.
3. Patients suffering from Type I Diabetes Mellitus
4. Patients with reduced daily caloric intake at baseline (≤ 2000 kcal/day) or malnutrition.
5. Patients who are already on a consistent and rigorous exercise regimen.
6. Gastrointestinal dysfunction requiring parental nutrition.
7. History of functional kidney transplant < 6 months prior to study entry.
8. Anticipated live donor kidney transplant over study duration.
9. Patients taking anti-inflammatory medication except aspirin < 325mg/day over the past 30 days.
10. Patients taking Vitamin E supplements > 60 IU/day, vitamin C > 500mg/day over the past 30days.
11. Patients taking any prednisone therapy.
12. Hospital admission within the last 30 days.
13. On experimental drug protocols.
14. Significant cardiac or vascular disease (symptomatic disease; CV event(s) within the last year; significant occlusive atherosclerotic disease or ischemic disease on non-invasive or invasive diagnostic procedures).
15. Significant physical disability or immobility (joint disease, joint replacement, muscular disorders).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2007-12; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
a statistically significant decrease in plasma F2-isoprostanes, a specific oxidative stress marker | 3 months
a statistically significant decrease in hs-CRP, a specific inflammatory marker | 3 months

SECONDARY OUTCOMES:
significant changes in additional markers of oxidative stress and inflammation | 3 months
significant changes in insulin resistance and adipocytokines | 3 months
a significant improvement in endothelial function as measured by brachial artery FMD | 3 months
a significant improvement in quality of life scores | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Alp Ikizler, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States